CLINICAL TRIAL: NCT07356765
Title: Berberine in Treating Negative Symptoms of Schizophrenia: Clinical Efficacy and Mechanisms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBR-SCH-NS
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Negative Symptoms of Schizophrenia
Keywords: schizophrenia; Negative Symptoms of Schizophrenia; berberine; Clinical efficacy; Mechanism of action
MeSH Terms: conditions — Schizophrenia | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- berberine group (Experimental)
  Interventions: Drug: Berberine
- control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berberine — Berberine 300 mg by mouth each dose# three times a day# plus any stable antipsychotic drug
  Other Names: stable antipsychotic
  Arms: berberine group
Drug: Placebo — The placebo were matched to Berberine in shape, smell and colour and tablets were sealed in identical bottles
  Other Names: stable antipsychotic
  Arms: control group

SUMMARY:
"Negative" symptoms are a major challenge for people with schizophrenia (SZ) and are a key reason why they struggle with everyday functioning. While current medications work well for the "positive" symptoms (like hallucinations or delusions), they aren't very effective at improving these "negative" symptoms, which include things like a lack of motivation or emotion. This study plans to conduct a large, randomized, double-blind, placebo-controlled trial to see if a compound called berberine (BBR) can safely and effectively improve these negative symptoms in SZ. The investigators will also examine how BBR affects gut bacteria, their byproducts in stool, and levels of general inflammation in the body. By looking at these different biological markers before and after BBR treatment, the investigators aim to understand how BBR influences negative symptoms and identify its main targets for improvement. This could lead to new ways to treat negative symptoms in schizophrenia in the future.

DETAILED DESCRIPTION:
The investigators will enroll at least 120 patients with schizophrenia (SZ) meeting the inclusion criteria, randomized 1:1 to either the experimental group receiving antipsychotic medication plus berberine (BBR) or the control group receiving antipsychotic medication plus placebo, for a clinical intervention of 12 weeks. The primary outcome measures will be the change in the Negative Symptom Scale (SANS) total score and the log50 result of the skin nicotine test throughout the 12-week period. Secondary outcome measures include the Positive and Negative Syndrome Scale (PANSS), the Clinical Global Impression scale (CGI), the Calgary Depression Scale for Schizophrenia (CDSS), the Global Assessment of Functioning (GAF), the Extrapyramidal Symptom Rating Scale, and cognitive assessments (MATRICS Consensus Cognitive Battery - MCCB). Other study indicators will involve the collection of sociodemographic and general clinical data. Blood and stool samples will be collected at pre-intervention (baseline), at 12 weeks of intervention, or at study termination. For safety assessments, participants' vital signs will be monitored at baseline, 4 weeks, 8 weeks, and 12 weeks, along with physical parameters (height, weight, blood pressure). Laboratory investigations will include complete blood count, comprehensive biochemical panel, and electrocardiogram (ECG). The Treatment Emergent Symptom Scale (TESS) will be used to assess drug side effects, and any adverse events will be recorded. Ultimately, the collected data will be used to investigate the clinical efficacy and safety of BBR on negative symptoms in SZ, its impact on the gut microbiota and their metabolic small molecules, its effect on peripheral blood inflammatory factors in SZ patients, and the longitudinal and cross-sectional correlations between gut microbiota and their metabolic small molecules, blood parameters, and negative symptoms in SZ patients under BBR treatment. This will facilitate the identification of early predictive biomarkers for BBR efficacy and key gut microbiota targets responsible for improving negative symptoms in SZ.

ELIGIBILITY:
Inclusion Criteria:

* Subjects met the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The diagnosis was confirmed by two psychiatrists who interviewed enrolled patients using the Structured Clinical Interview for DSM-5 Disorders, Clinician Version (SCID-5-CV).
* Age between 18 and 60 years, inclusive.
* Gender: Not restricted.
* Ethnicity: Han Chinese.
* Subjects were receiving a stable dose of antipsychotic medication for at least 3 months prior to enrollment and had no dose adjustments in the month preceding enrollment.
* Subjects exhibited significant negative symptoms, defined as: A total score of ≤ 70 on the Positive and Negative Syndrome Scale (PANSS). Scores of ≤ 4 on the PANSS items for delusions, conceptual disorganization, hallucinations, and excitement. A score > 0 on the Negative Symptom Subscale-Positive Symptom Subscale.
* The patient or their legal representative provided informed consent and signed the informed consent form agreeing to participate in the study.

Exclusion Criteria:

* Individuals meeting DSM-5 criteria for other psychiatric disorders.
* Current severe neurological disease, uncontrolled metabolic disease, infectious disease, or autoimmune disease.
* History of gastrointestinal surgery.
* Use of antibiotics, other immunomodulatory agents, hormones, microecological agents, or probiotic medications within the past 1 month.
* Allergy to BBR (if "BBR" is a known abbreviation, otherwise it should be spelled out or defined).
* Receipt of physical therapies such as electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) within the past 1 month.
* Individuals with hemolytic anemia and glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Pregnant or lactating females.
* Any factor that would prevent the participant from providing informed consent or participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in the total score of the Scale for Assessment of Negative Symptoms (SANS) | Baseline, week4, week8, week12
  The Scale for Assessment of Negative Symptoms (SANS) is a clinician-rated observational scale developed by American neuropsychiatrist Nancy C. Andreasen to assess negative symptoms in schizophrenia. The scale includes categories such as alogia (poverty of speech), blunted affect, avolition, anhedonia/asociality, and attention impairment, with a focus on evaluating the patient's deficit symptoms of mental activity. Changes in the total SANS score will, to a certain extent, reflect changes in the severity of the subject's negative symptoms.
log50 of the cutaneous niacin flush | Baseline, week4, week8, week12
  In this study, the Skin Flush Meter will be utilized for the first time to quantify the attenuation of the niacin flush response, serving as an objective assessment tool for negative symptoms in schizophrenia (SZ). Building upon a pre-existing image library of niacin flush responses from a previous cohort, the research team from our collaborating unit has developed a niacin predictor device. This device largely preserves the observational steps of the original method. Based on this, previously manual simple scoring has been replaced with artificial intelligence (AI) for processing large volumes of color images. It compares pre- and post-niacin color differences in the skin, extracts variables for erythema intensity, and precisely calculates the area of irregular redness. By integrating the temporal dimension, it further achieves quantification and refinement with second-level resolution.

SECONDARY OUTCOMES:
Cognitive Function | Baseline, week4, week8, week12
  All participants underwent cognitive function assessment based on the MATRICS Consensus Cognitive Battery (MCCB). There are 9 subtests, which mainly assess 7 cognitive domains, including information processing speed, attention/alertness, Working memory, word learning, visual memory, reasoning and problem solving, and social cognition. After the evaluation is completed, the MCCB rough score is converted into the total score T score obtained after correction for age, gender, years of education, and untreated period. The T score is then converted into a defect score, with T scores ≥ 40, 35-39, 30-34, 25-29, 20-24, and ≤ 19 corresponding to defect scores 0, 1, 2, 3, 4, and 5, respectively. Among them, 1 represents mild defects, 2 represents mild to moderate defects, 3 represents moderate defects, 4 represents moderate to severe defects, and 5 represents severe defects. In this study, a defect score of ≥ 3 was used as the boundary for significant cognitive impairment.
Psychiatric Symptoms | Baseline, week4, week8, week12
  The psychiatric symptoms of schizophrenia were assessed in all enrolled patients using the Positive and Negative Syndrome Scale (PANSS). The PANSS is a 30-item clinician-rated scale yielding a total score ranging from 30 (least symptomatic) to 210 (symptomatic), where higher scores indicate more severe psychopathology.
Clinical efficacy | Baseline, week4, week8, week12
  The Clinical Global Impression (CGI) scale is a standardized tool used to assess the severity of a patient's illness and the effectiveness of treatment. The CGI employs a 1 to 7 point graded rating scale, with two subscales: Clinical Global Impression of Severity (CGI-S) and Clinical Global Impression of Improvement (CGI-I). Higher CGI-S scores indicate greater illness severity. CGI-I is calculated as the difference between post-treatment and pre-treatment assessments; a higher score signifies more significant illness improvement.
Depressive Symptoms | Baseline, week4, week8, week12
  The Calgary Depression Scale for Schizophrenia (CDSS) is primarily utilized to evaluate depressive symptomatology in patients with schizophrenia. The scale consists of 9 structured items that assess: depressive mood, despair, self-deprecation, delusions of guilt, pathological guilt, diurnal variation (morning depression), early morning awakening, suicidal ideation, and observed depressive signs. Each item is rated on a 0-3 point scale, where higher scores signify increased symptom severity.
Functional capacity | Baseline, week4, week8, week12
  The Global Assessment of Functioning (GAF) Scale for individuals with schizophrenia is a specialized instrument for evaluating their functional capacity. Its purpose is to comprehensively assess the patient's functional performance in various significant life areas, such as social, occupational, and psychological functioning, as well as activities of daily living. The scale's scoring ranges from 0-100:
  A score of ≥ 71: Suggests generally normal social functioning, enabling regular engagement in work, study, and social activities.
  A score of 51-70: Implies mild impairment in social functioning, possibly characterized by diminished social interactions or reduced responsibility.
  A score of 31-50: Denotes significant impairment in social functioning, necessitating ongoing supervision or supportive assistance for daily living.
  A score of ≤ 30: Signifies severe impairment in social functioning, requiring professional therapeutic or custodial care.
Changes of CRP | Baseline, week12
  The concentration of C-reactive protein (CRP) is measured in venous blood. CRP is an acute-phase reactant protein synthesized by the liver, primarily functioning to recognize and clear pathogens or damaged cells. It plays a crucial role in inflammatory responses, infection surveillance, and disease monitoring.
Fecal 16S rRNA sequencing | Baseline, week12
  Fresh morning stool samples were collected from subjects at baseline, 12 weeks, or study termination using a 5ml sterile, sealed stool collection kit. Care was taken to collect from the center of the sample, avoiding contact with the external environment to prevent contamination. Within 15 minutes of collection, samples were divided into two 2ml EP tubes and stored at -80°C for fecal 16S rRNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, China